CLINICAL TRIAL: NCT06524115
Title: Optimization of a Photoretinoscopy Method for Determining the Objective Refraction of Children With a Smartphone/add-on Device in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: WS10364
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Photorefraction prototype device (Experimental): - Photoretinoscopic images without cycloplegia
  Interventions: Device: Comparator device, Closed-field autorefractometer without cycloplegia; Other: Distance visual acuity check using objective refraction without cycloplegia; Device: Comparator device, Closed-field autorefractometer with cycloplegia; Other: Distance visual acuity check using objective refraction with cycloplegia

INTERVENTIONS:
Device: Comparator device, Closed-field autorefractometer without cycloplegia — Objective refraction without cycloplegia
Other: Distance visual acuity check using objective refraction without cycloplegia — Distance visual acuity is checked, using objective refraction without cycloplegia
Device: Comparator device, Closed-field autorefractometer with cycloplegia — Objective refraction with cycloplegia
Other: Distance visual acuity check using objective refraction with cycloplegia — Distance visual acuity is checked, using objective refraction with cycloplegia

SUMMARY:
The objective is to compare the refractive parameters of the photorefraction prototype device without cycloplegia with the refractive parameters of reference device, an autorefractometer with and without cycloplegia.

DETAILED DESCRIPTION:
A single visit will be necessary. After informed consent, and checking of the inclusion and exclusion criteria, investigators will perform measurements with an autorefractometer and with the photorefraction prototype device without cycloplegia followed by an objective refraction with an autorefractometer under cyclopegia.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary, willing to follow the protocol, able to read and understand the information form and give free and informed consent (for parents/guardian of children subjects) and assent (for subjects aged 6-12 years old
* At least 6 years old and up to 12 years old at time of informed consent and assent
* Average of the equivalent sphere(Sph+Cyl/2) of both eye included in the interval [-10.00, +8.00]
* Cylindrical refractive error between 0 and 4.00 D on both eyes
* Corrected binocular visual acuity in distance vision at least 6/9

Exclusion Criteria:

* Incapable of expressing consent
* All categories of persons particularly protected by law
* Subject in another study which might have an influence on vision or interfere with study assessment
* Less than 6 years old, or 13 years old or above at time of informed consent and assent
* Amblyopia, Cataract, Strabismus.
* Aphakic or pseudophakic (intraocular implant)
* Reported severe eye disease involving loss of visual field as in glaucoma, involving loss of acuity and severe discomfort in low or overly bright environments as in retinitis pigmentosa or reported and treated dry eye.
* Self-reported neurological deficits, including a history of epileptic pathology or sensory-motor coordination disorders, vestibular or cerebellar pathology (e.g., balance disorders, nystagmus)
* Any previous ocular surgery, which might have an influence on vision or interfere with study assessments (e.g. iridectomy, refractive surgery…),
* Any myopia control solutions that could affect refractive status of the eye (e.g. Atropine eye drops, Orthokeratology)

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Objective refractive error | One day (all measurements are taken during the single visit)
  The refractive error is collected in sphere power (D), cylinder power (D) and cylinder axis (°) and converted in equivalent sphere, J0, J45 (power vector in D)

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Kumar, Principal Investigator — Sankara Nethralaya, Unit of Medical Research Foundation
Locations (1):
- Sankara Nethralaya, Unit of Medical Research Foundation, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No